CLINICAL TRIAL: NCT04121871
Title: Formulation Development and In-Vitro Studies of Efficacy of Botanical Extracts Against Candida Auris
Brief Title: Molecular Characterization of Candida Auris
Acronym: OC
Status: Completed | Type: Observational
Sponsor: Islamia University of Bahawalpur (Other)
Responsible Party: Principal Investigator, Jafir Hussain Shirazi, Principal Investigator, Islamia University of Bahawalpur
Other Study IDs: Oral Fungal Infection
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Oral Fungal Infection
Keywords: Candida auris; Oral Fungal Infection; Candidiasis
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Clinical oral swab samples from infected patients will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Not required

SUMMARY:
Candida auris is emerging fungal opportunistic pathogen in developing countries. Much studies has been conducted on Candida albicans. there was a dire need to investigate this alarming threat. Our hypothesis is that by recording the patients diagnosed with oropharygneal candidiasis and collecting clinical swab samples from these patients will be fruitful if microbiological isolation, identification and molecular characterization will be done. So this is the first study on C. auris in south punjab, Pakistan. Aim of this study is to collect epidemiological data of C. auris.

ELIGIBILITY:
Inclusion Criteria:

* Pre-diagnosed Patients of both gender from pre-selected localities

Exclusion Criteria:

* Healthy individuals or individuals having no oral fungal infection individuals above 100 years of age

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals are equally eligible to be selected in the study
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of C. auris | From November 15, 2019 to February 29, 2020
  patients from selected localities will be recorded along with total patients in that category, prevalence will be calculated on the record collected from specified duration of study
Seasonality of C. auris infection | From November 15, 2019 to February 29, 2020
  Number of patients recorded during different months will be the source of calculation of seasonality index of the C. auris infection
Drug susceptibility | From November 15, 2019 to February 29, 2020
  Antifungal drug discs will be used for assessing the antfungal drugs susceptibility

CONTACTS AND LOCATIONS:
Overall Officials: Jafi H Shirazi, M.Phil, Principal Investigator — The Islamia University of Bahawalpur
Locations (2):
- Pakistan (2):
  - Bahawal Victoria Hospital Bahawalpur, Bahawalpur, Punjab Province
  - Civil Hospital Jhangi Wala Road Bahawalpur, Bahawalpur, Punjab Province

IPD SHARING:
Plan to Share IPD: No
Individual privacy is prime important, hence data will not be shared